CLINICAL TRIAL: NCT05689346
Title: High Tone Power Therapy Improves Balance and Quality of Life in Hemiparetic Cerebral Palsy Children: A Randomized, Double Blind, Placebo-controlled Trial
Brief Title: High Tone Power Therapy for Hemiparetic Cerebral Palsy Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Shafiek Mustafa Saleh, assistance professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: high tone therapy for CP.
Record Dates: First submitted 2023-01-08; First posted 2023-01-19 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Hemiparetic Cerebral Palsy Children

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): study group will receive high tone power therapy
  Interventions: Device: high tone power therapy
- control group (Active Comparator): children in the contol group will recieve traditional treatment for improving balance.
  Interventions: Other: traditional physical therapy exercises

INTERVENTIONS:
Device: high tone power therapy — high tone power therapy
  Arms: study group
Other: traditional physical therapy exercises — traditional physical therapy exercises for improving balance
  Arms: control group

SUMMARY:
Balance reactions and postural control are inadequate in children with CP which affect their daily living activities. So, different treatment modalities have been used to improve balance for cerebral palsy children. Recently, High tone power therapy is a new quantum leap in the field of electro therapy that can be used to stimulate nerves and muscles, so this randomized controlled study will be conducted to investigate the effect of high tone power therapy on balance and quality of life in hemiparetic cerebral palsy children.

ELIGIBILITY:
Inclusion criteria:

* Age ranged from 6 to 8 years.
* Height not less than one meter.
* Their spasticity will range from 1 to 1+ according to the Modified Ashworth Scale.
* Children have normal flexibility of the lower back muscles as adequate flexibility with normal muscle length is essential for proper joint function and efficient movement.
* Exclusion criteria:
* Children will not follow instructions.
* Children with any cardiopulmonary problems, attitude and psychiatric disorders, length discrepancy; and seizures.
* Tightness of the hip flexors.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
balance assessment | change from base line at 4 weeks.
  biodex balance system will be used to assess the dynamic balance: Before the evaluation procedures all children will be given an explanatory session to be aware about the different test steps, also the support rails and biofeedback display screen will be adjusted for each child to ensure comfort and safety during the test procedure, then each child will be trained 1 min for adaptation to the machine. During the test, children will be instructed to stand on the platform in the most comfortable posture, and maintain their visual level by focusing straight ahead on the monitor. The platform will be unlocked and children will be allowed to adjust their foot placement until a comfortable standing position will be achieved while they simultaneously maintained a moving pointer at the center point on the monitor and children will be encouraged to maintain the moving pointer at the center point throughout the test.

SECONDARY OUTCOMES:
quality of life assessment | change from base line at 4 weeks.
  The Pediatric Quality of Life Inventory (PedsQL) is a questionnaire assessment tool used to evaluate HRQOL in children. It is composed of 23 items that gauge function in the following four areas: physical (eight items), emotional (five items), social (five items), and school (five items). Patients report their function using a 5-point Likert scale ranging from 0 to 4. These responses are reverse scored and linearly transformed to a 0 to 100 scale, with a higher score indicating a higher QOL.